CLINICAL TRIAL: NCT03883984
Title: Cysteamine for Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Hershey-101
Record Dates: First submitted 2018-12-27; First posted 2019-03-21 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Cysteamine

STUDY DESIGN:
Intervention Model Description: 1:1 randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cysteamine (Experimental): Cysteamine Bitartrate plus standard asthma care
  Interventions: Drug: Cysteamine Bitartrate
- Placebo Oral Tablet (Placebo Comparator): Placebo plus standard asthma care
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Cysteamine Bitartrate — Cysteamine bitartrate administered four times per day (QID) for 8 weeks. 125mg tablet QID.
  Arms: Cysteamine
Drug: Placebo Oral Tablet — Placebo administered for 8 weeks. 125mg tablet QID.
  Arms: Placebo Oral Tablet

SUMMARY:
The purpose of this study is to see if a medicine called Cysteamine, given along with standard asthma care, will improve asthma symptoms and lung function.

DETAILED DESCRIPTION:
Asthma affects 25.7 million people in the US. Many people report symptoms despite taking high-doses of inhaled asthma medications. This difficult-to-treat group accounts for more than 50% of asthma related healthcare visits and hospitalizations. The purpose of this study is to see if a medicine called Cysteamine, given along with standard asthma care, will improve asthma symptoms and lung function.

This study is a double-blind, placebo-controlled, randomized trial of cysteamine. A placebo arm will be included to determine the comparative effectiveness of cysteamine in this population. Eligible participants will be assessed 1, 4 and 8 weeks post randomization and followed for an additional 4 weeks post treatment.

In order to enroll in this study, participants must be between the ages of 18-45 and have uncontrolled asthma.

This study will include 4 visits and weekly phone calls, and will be in the study for 3-4 months.

During the treatment period, participants will be placed in one of two treatment groups:

* Cysteamine
* Placebo

Participants will not be able to choose which group they are assigned. This assignment is random and by chance, much like flipping a coin. Participants will not know if they are receiving Cysteamine or placebo. Investigators will compare the study results between the participants of each group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥ 18 years and ≤ 45 years
* Provision of written informed consent
* Asthma currently treated with moderate-high doses of Inhaled Corticosteroids (ICS) per the National Asthma Education and Prevention Program (NAEPP) guidelines by self-report
* Evidence of hypersensitivity to environmental allergens, with at least one of the following:
* Elevated serum IgE
* Positive allergy skin prick testing to at least 1 allergen.
* Evidence of allergic rhinitis by physical exam or by medical history.
* Peripheral blood eosinophils ≥150 cells/µl obtained at screening visit.
* Asthma Severity Score indicating Moderate to Severe Impairment based on EPR-3 classification guidelines
* > 1 utilization for treatment of asthma exacerbation including prescription of oral or intravenous steroids (urgent care, emergency department visit, or hospitalization for asthma) in the past 12 months
* Negative urine pregnancy test for females of child bearing potential and use of contraception throughout the study.

Exclusion Criteria:

* Diagnosis of chronic lung disease other than asthma
* Have received biologic therapy (e.g., anti-IgE, anti-IL-4, anti-IL-5) within 6 months of study entry.
* Diagnosis of chronic disease other than asthma requiring daily steroids or immunosuppressive agents
* History of a heart attack or severe chronic heart disease
* Current smoking or previous history within 1 year
* Transplant patient
* IBD, Crohn's
* History of ulcer, gastric esophageal reflux (GERD) or chronic peptic ulcer disease
* Pregnant or planning to become pregnant
* Breastfeeding
* History of severe allergic or anaphylactic reactions to medications
* Grade 2-4 Abnormal Laboratory Results (hemoglobin, WBC, lymphocytes, platelets, sodium, potassium, glucose, BUN, creatinine, calcium, albumin, total protein, alkaline phosphate, AST, ALT, and bilirubin), see table 7.4.1.2a and 7.4.1.2b.
* Grade 3-4 Abnormal Eosinophils and Neutrophils, see table 7.4.1.2a.
* Evidence of papilledema, or history of pseudotumor cerebri
* History of persistent headaches
* Allergic reaction to cysteamine or penicillamine
* Serious medical condition that, in the opinion of the Study Investigator, would interfere with the ability of the patient to complete the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Change in the Asthma Symptom Severity Score | Baseline (Pre-Treatment), V1 (4 weeks), V2 (8 weeks), Study End (4 weeks post-treatment, Follow-up Phone Call)
  Asthma symptom severity score will be classified using the Expert Panel Report 3 (EPR-3) criteria for untreated asthma. The level of impairment is based on the most severe indication of the following criteria: 1. Symptoms, 2. Nighttime awakenings, 3. Short-Acting Beta Agonist (SABA) use for symptom control, 4. Interference with normal activity, and 5. Lung Function.

SECONDARY OUTCOMES:
Number of Days with Albuterol Use Over Time | Baseline (Pre-Treatment), V1 (4 weeks), V2 (8 weeks), Study End (4 weeks post-treatment, Follow-up Phone Call)
  Albuterol is a bronchodilator used as a rescue medication for treatment of asthma symptoms.
Change in Inflammation in TH2 cells Over Time | Baseline (Pre-Treatment), V1 (4 weeks), V2 (8 weeks, End Treatment)
  Inflammation as measured by T Helper Type 2 (TH2) cells in peripheral blood.
Spirometry Measurement: Forced Expiratory Volume in 1 second (FEV1) Over Time | Baseline (Pre-Treatment), V1 (4 weeks), V2 (8 weeks, End Treatment)
  FEV1 is the amount of air exhaled in 1 second during spirometry. This is used as a measurement of asthma severity.
Peak Flow Measurement: Forced Expiratory Volume in 1 second (FEV1) Over Time | Baseline (Pre-Treatment), V1 (4 weeks), V2 (8 weeks), Study End (4 weeks post-treatment, Follow-up Phone Call)
  FEV1 will be obtained by peak flow measurement. This will be used as a measurement in asthma severity.
Peak Flow Measurement: Peak Expiratory Flow (PEF) Over Time | Baseline (Pre-Treatment), V1 (4 weeks), V2 (8 weeks), Study End (4 weeks post-treatment, Follow-up Phone Call)
  PEF will be obtained by peak flow measurement. This will be used as a measurement in asthma severity.
Change in Asthma Quality of Life Questionnaire (miniAQLQ) scores Over Time | Baseline to Visit 2 (8 weeks)
  The miniAQLQ will be used to measure the impact that asthma has on participants quality of life. The miniAQLQ will ask questions in the following domains: symptoms, activity limitations, emotional function, and environmental stimuli. There are 15 questions, each with a 7-point scale. An answer of 1 on a question represents the greatest impairment possible and a 7 represents the least impairment. Individual questions are equally weighted. The overall miniAQLQ score is the mean of the responses to each of the 15 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Gurjit K Khurana Hershey, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States